CLINICAL TRIAL: NCT04820556
Title: The Development of Preventive Methods for Chronic Noncommunicable Diseases Based on Modulation of Gut Microbiota Composition and Function
Brief Title: Gut Microbiota in Chronic Noncommunicable Diseases
Status: Completed | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: Center for Strategic Planning and Management of Biomedical Health Risks of the Federal Biomedical Agency (Unknown)
Responsible Party: Principal Investigator, Anastasia Kaburova, junior researcher, National Medical Research Center for Therapy and Preventive Medicine
Other Study IDs: 3162021
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Arterial Hypertension; Atherosclerosis Occlusive Disease; Heart Failure With Preserved Ejection Fraction; Heart Failure With Reduced Ejection Fraction; Diabetes Mellitus, Type 2; Obstructive Pulmonary Disease; Asthma; Nonalcoholic Fatty Liver Disease
Keywords: chronic noncommunicable diseases; gut permeability; inflammation; gut microbiota
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Lung Diseases, Obstructive; Asthma; Non-alcoholic Fatty Liver Disease; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum, plasma, stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Arterial hypertension
- Atherosclerosis occlusive disease
- Heart failure with preserved ejection fraction
- Heart failure with reduced ejection fraction
- Diabetes mellitus, type 2
- Chronic obstructive pulmonary disease and asthma
- Nonalcoholic fatty liver disease
- Control group

SUMMARY:
It is an observational study in patients with chronic noncommunicable diseases (i.e. cardiovascular diseases, diabetes mellitus, non-alcoholic fatty liver disease, chronic obstructive pulmonary disease and asthma ) and control group with no signs of these conditions. The study has a prospective part planned for 2021 and a retrospective part which includes the patients enrolled between 2018-2020. The aim of the study is to investigate gut microbiota composition, its metabolites, levels of inflammatory and other markers of the disease in prospective groups (arterial hypertension, type 2 diabetes mellitus, chronic obstructive pulmonary disease, asthma, non-alcoholic fatty liver disease and control patients) as well as in retrospective groups (chronic heart failure with preserved and reduced ejection fraction, obstructive atherosclerosis of any vascular bed, arterial hypertension, type 2 diabetes mellitus, chronic obstructive pulmonary disease, asthma, non-alcoholic fatty liver disease, and control patients). Also we are planning to investigate the association between gut microbiota composition and its metabolites, levels of inflammatory and other markers of the disease in retrospective and prospective groups.

ELIGIBILITY:
Criteria for groups with arterial hypertension, chronic obstructive pulmonary disease (COPD), asthma, type 2 diabetes mellitus and nonalcoholic fatty liver disease (NAFLD) (both prospective and retrospective)

Inclusion criteria:

All mentioned groups:

* Men and women aged ≥ 18 and <80
* Signed informed consent form

Group of arterial hypertention (inclusion criteria):

1. No current treatment of hypertension
2. Systolic blood pressure <180 mm Hg and diastolic blood pressure <110 mm Hg
3. No clinical signs of other cardiovascular diseases

Group of COPD and asthma (inclusion criteria)

1. Medical records, confirming COPD or asthma
2. Regular stable treatment of COPD, asthma or any chronic disease for ≥ 4 weeks before the enrollment. If inhaled corticosteroids are being used, regular treatment is required for ≥12 weeks.
3. Absence of acute exacerbations of COPD, asthma or any concomitant diseases 4 weeks before the enrollment
4. No use of genetically engineered biological drugs
5. For patients with COPD after inhalation of salbutamol (400 mcg) the ratio FEV1/FVC is less than 0,70

Group of type 2 diabetes mellitus (inclusion criteria)

1. Confirmed type 2 diabetes mellitus
2. Stable glucose lowering treatment for ≥ 1 month
3. No systemic corticosteroid treatment 4 weeks before the enrollment

Group of NAFLD (inclusion criteria)

1. Ultrasound criteria of non-alcoholic fatty liver disease or
2. Confirmed non-alcoholic fatty liver disease using FibroMax test

Control group inclusion criteria

1. Men and women aged ≥ 18 and <80 years
2. Signed informed consent form

Control group for arterial hypertension (inclusion criteria):

1. No history of cardiovascular diseases, COPD or asthma

Control group for COPD and asthma (inclusion criteria):

1. No history of diabetes mellitus, NAFLD, COPD and asthma

Exclusion criteria for all groups

1. Age < 18 years and ≥80 years
2. Denial of further participation
3. Obesity with BMI≥40 kg/m2
4. History of organ transplantion
5. Psychiatric disorder, limiting participation in the study
6. Acute infections
7. Exacerbation of chronic infection 2 weeks before the enrollment
8. Cancer with no radical treatment
9. Pregnancy and lactation
10. Alcohol and drug addition
11. Chronic kidney disease with GFR <30 ml/min/1.73m2
12. Systemic autoimmune diseases
13. Inflammatory bowel disease
14. Antimicrobial and probiotic treatment 3 months before the enrollment

Additional exclusion criteria adjusted for each group

Group of arterial hypertension (exclusion criteria):

1. Ischemic heart disease (angina pectoris, myocardial infarction), cerebrovascular disease (stroke, transient ischemic attack), occlusive peripheral arterial disease, revascularization of any vascular bed.
2. Cardiomyopathies
3. Symptomatic arterial hypertension
4. Diabetes mellitus
5. Signs of previous myocardial infarction on ECG
6. Arrhythmias (parohysmal arrhythmias, atrial fibrillation, sinoatrial block, atrioventricular block grade II-III)
7. Signs of current myocardial ischemia on ECG
8. Decompensated heart failure

Group of COPD and asthma (exclusion criteria):

1. Exacerbation of COPD or asthma 3 months before the enrollment which required antibiotic treatment or systemic corticosteroids.

   Group of type 2 diabetes mellitus (exclusion criteria):
2. Type 1 diabetes mellitus and other specific types of diabetes
3. Severe microangiopathy: proliferative and terminal stage of diabetic retinopathy, chronic kidney disease (GFR < 30 ml/min/1,73 m2) for patients with type 2 diabetes
4. The history of moderate, severe and very severe COPD
5. The history of moderate or severe asthma
6. Vegetarians or vegans

Group of non-alcoholic fatty liver disease (exclusion criteria):

1. Chronic liver diseases except NAFLD
2. The history of moderate, severe and very severe COPD
3. The history of moderate or severe asthma
4. Vegetarians or vegans
5. Diabetes mellitus

Criteria for groups of heart failure and obstructive atherosclerosis (retrospective)

Inclusion criteria for HF-pEF group:

1. Men and women aged ≥ 18 and <80 years
2. Signs and symptoms of heart failure
3. Left ventricular diastolic dysfunction
4. Left ventricular ejection fraction ≥50%
5. NT-pro BNP >125 pg/ml
6. Signed study informed consent form

Inclusion criteria for HF-rEF group:

1. Men and women aged ≥ 35 and <80 years
2. Signs and symptoms of heart failure
3. Left ventricular ejection fraction <50%
4. Signed study informed consent form

Inclusion criteria for obstructive atherosclerosis group:

1. Men and women aged ≥ 35 and <80 years
2. Symptoms and signs of obstructive atherosclerosis of any vascular bed:

   1. Ischemic heart disease or
   2. Revascularization of coronary, renal, brachiocephalic or lower extremity arteries or
   3. carotid endarterectomy or
   4. chronic lower extremity ischemia or
   5. history of myocardial infarction, stroke, transient ischemic attack or
   6. renovascular AH
   7. atherosclerotic aorta aneurysm
3. Signed study informed consent form

Inclusion criteria for control group for HF-pEF, HF-rEF and obstructive atherosclerosis

1. Men and women aged ≥ 18 and <80 years.
2. No signs or symptoms of chronic heart failure
3. No signs of left ventricular diastolic dysfunction
4. No history, signs or symptoms of obstructive atherosclerosis of any vascular bed
5. Signed study informed consent form

Exclusion criteria for groups with HF-pEF, HF-rEF and obstructive atherosclerosis:

1. Age <18 and ≥80 years.
2. Refuse to sign study informed consent form
3. Body mass index ≥35 kg/m2
4. Chronic kidney disease with GFR <30 ml/min/1,73 m2
5. Current smoking
6. Moderate or severe COPD
7. Moderate or severe asthma
8. Acute infections or exacerbation of chronic infections 2 weeks prior to study enrollment
9. History of allergic reactions to gadolinium contrast
10. Hypertrophic cardiomyopathy, dilated cardiomyopathy, restrictive cardiomyopathy: primary, amyloidosis, glycogen storage diseases, hemochromatosis, sarcoidosis, drug induced cardiomyopathy, radiation heart disease, constrictive pericarditis).
11. Connective tissue disease
12. Cancer with no radical treatment
13. Pregnancy or lactation
14. Inflammatory bowel disease
15. Use of antimicrobial agents, probiotics or systemic corticosteroids 3 months before the enrollment

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic noncommunicable diseases including cardiovascular diseases, type 2 diabetes mellitus, nonalcoholic fatty liver disease, chronic obstructive pulmonary disease, asthma and control group
Sampling Method: Non-Probability Sample
Enrollment: 1084 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Significant (p<0,05) correlation (r>0,5) between abundance of Faecalibacterium genus and concentration of lipopolysaccharide | on enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - National Medical Research Center for Therapy and Preventive Medicine of the Ministry of Healthcare of the Russian Federation, Moscow
  - Centre for Strategic Planning and Management of Biomedical Health Risks of the Federal Medical Biological Agency, Moscow

IPD SHARING:
Plan to Share IPD: No